CLINICAL TRIAL: NCT02591108
Title: Quantitative Assessment of Train of Four Device for Patients Receiving Neuromuscular Blockade
Brief Title: Train of Four Motor Point Stimulation and Monitoring
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201501M61361
Record Dates: First submitted 2015-03-18; First posted 2015-10-29 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Observation of Neuromuscular Block
Keywords: train of four; neuromuscular blockade; surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Safety and Efficacy (Experimental): Parallel treatment; use of standard TOF peripheral Stimulator to Novel Train of Four Device
  Interventions: Device: Neuromuscular Block Aid; Device: Standard of Care: Microstim Plus
- Microstim (Active Comparator): A peripheral nerve stimulator, also known as a train-of-four monitor, is used to assess neuromuscular transmission when neuromuscular blocking agents (NMBAs) are given to block musculoskeletal activity. By assessing the depth of neuromuscular blockade, peripheral nerve stimulation/monitoring can ensure proper medication dosing and thus decrease the incidence of side effects. Peripheral nerve stimulation is most commonly used for ongoing monitoring in the intensive care unit (ICU).
  Interventions: Device: Neuromuscular Block Aid; Device: Standard of Care: Microstim Plus

INTERVENTIONS:
Device: Neuromuscular Block Aid — Neuromuscular Block Aid, is a quantitative mechansim for collecting the the train-of-four and can be kept in an electronic medical record, also known as a train-of-four monitor, is used to assess neuromuscular transmission when neuromuscular blocking agents (NMBAs) are given to block musculoskeletal activity. By assessing the depth of neuromuscular blockade, peripheral nerve stimulation/monitoring can ensure proper medication dosing and thus decrease the incidence of side effects. Peripheral nerve stimulation is most commonly used for ongoing monitoring in the intensive care unit (ICU).
  Other Names: Peripheral Nerve Stimulator - Train of Four Monitoring
Device: Standard of Care: Microstim Plus — A peripheral nerve stimulator, also known as a train-of-four monitor, is used to assess neuromuscular transmission when neuromuscular blocking agents (NMBAs) are given to block musculoskeletal activity. By assessing the depth of neuromuscular blockade, peripheral nerve stimulation/monitoring can ensure proper medication dosing and thus decrease the incidence of side effects. Peripheral nerve stimulation is most commonly used for ongoing monitoring in the intensive care unit (ICU).

SUMMARY:
The assessment of neuromuscular blockage is common practice in the operating room, in which such agents are employed. Still today, the use of simple hand held stimulators and visual monitoring of these responses are the norm. The investigators want to study the potential for employing a non-invasive quantitative device with built in sensors that will hopefully accurately determine the degree of neuromuscular blockade. This system utilizes commonly employed train of four (TOF) electrical stimulation pulses, an incorporated force sensor and an automated detection system. This system will not only utilized pre-blockade, but also throughout an entire surgical procedure and during reversal therapy. For comparisons, the investigators will use both the prototype device and a standard hand held TOF for the assessment of neuromuscular blockage. In other words, the planned protocol will involve testing the effectiveness and accuracy of the device concurrently with peripheral nerve stimulation, during a procedure as is done for the current standard of care. All protocols will be carried out under the direct guidance and supervision of anesthesiologists and/or nurse anesthetists.

DETAILED DESCRIPTION:
Project Summary:

In this study the investigators propose to evaluate a train of four (TOF) stimulator that assess the neuromuscular junction of a patient under anesthesia. The goal of this project is to evaluate a novel device in comparison to the standard of care with a hand held stimulator.

Background and Significance:

The assessment of neuromuscular blockage is common practice in the operating room, in which such agents are employed. Still today, the use of simple hand held stimulators and visual monitoring of these responses are the norm. The investigators now want to study the potential for employing a non-invasive quantitative device with built in sensors that will hopefully accurately determine the degree of neuromuscular blockade. This system utilizes commonly employed train of four (TOF) electrical stimulation pulses, an incorporated force sensor and an automated detection system. This system will not only utilized pre-blockade, but also throughout an entire surgical procedure and during reversal therapy. For comparisons, we will use both the prototype device and a standard hand held TOF for the assessment of neuromuscular blockage.

In other words, the planned protocol will involve testing the effectiveness and accuracy of the device concurrently with peripheral nerve stimulation, during a procedure as is done for the current standard of care. All protocols will be carried out under the direct guidance and supervision of anesthesiologists and/or nurse anesthetists.

The procedure involves applying the device to a suitable anatomic location for train of four (TOF) stimulation/monitoring and then applying a small electrical pulse to stimulate the patient's motor point. The location for this stimulation has historically been on the patients forearm over the ulnar nerve area or on the patients face in the distribution of the facial nerve. The stimulation applied to these areas is equivalent to that applied in the current accepted standard of care. All responses measured by the device will be recorded electronically and compared to anesthesiologist's/nurse anesthetist's interpretation of the number of muscle twitches induced by peripheral motor point stimulation. These comparisons will be analyzed for correlation between number of muscle twitches and degree of force generation sensed by the device, with the aim of more accurately determining the degree of the patients neuromuscular blockade.

This device application and monitoring will be carried out on anesthetized surgical patients at different time points in the procedure, under the same conditions as the currently utilized peripheral nerve stimulators to judge neuromuscular transmission and anesthesia effectiveness. We will also use the system on other anatomical locations that may be easier to gain assess to under certain surgical procedures: e.g., on the bicep, quadriceps, or tibialis anterior muscles. Such locations have been described by anesthesiologists as viable options.

Pre and post-surgical care will be unchanged and follow current standard of care. The only change will be that alongside current peripheral nerve stimulation, our non-invasive TOF device will also be utilized for assessing the relative degree of neuromuscular blockage.

Currently, there is no clinically available device that is automated and records the TOF conducted the anesthesiologist and their staff. Developing a method for completed this assessment is expected to save the anesthesiologist's time and prevent human error and increase consistency.

This device and approach is similar to the muscle force system which we have employed to study patients with neuromuscular disorders at the University of Minnesota for over 20 years.

Specific Aims/Study Objectives:

The investigators hypothesize that the use of an advance TOF device with automated data storage and a unique user interface will demonstrate enhanced efficacy for monitoring neuromuscular blockade in patients. The investigators will continue to recruit subjects for this study until we have completed the study.

Research Design and Methods:

The study population will include female and male participants ranging from 18-80 years of age. The investigators are requesting a total of 400 participants in the study. After the investigators have collected data from these individuals they will analyze the data to determine the efficacy of the testing method. If the initial population size is extremely variable or does not allow the investigators to conduct a proper analysis, they will request additional subjects to make a conclusion on this device.

Subject will be identified by the anesthesiologist prior to surgery, consent will be obtained prior to surgical procedures. The information that will be collected from their medical records will include their age, height, weight, history of muscular disease i.e. myotonias, malignant hyperthermia, previous adverse reactions to anesthesia, complete anesthetic records from procedure. Data will be securely stored and locked in Mayo B172.

Data and Safety Monitoring Plan:

It is not anticipated that the use of this device will produce any side effects or emotional upset. The stopping rules of the study include any unexpected complications with the use of the TOF stimulator in the OR. The patient will be unconscious or sedated during monitoring.

Statistical Considerations:

Historically, FDA clinical trials have utilized anywhere from 100-400 patients for determining the relative safety and efficacy of a medical device or technology. The obtained data will be analyzed to determine such factors and could be utilized for FDA approval of a monitoring system for clinical use.

Direct comparison of the devices qualitative evaluation of scoring from the administering anesthesiologist will be used for the final analysis.

Data and Record Keeping:

The data will be recorded by Dr. Michael Loushin, Dr. Paul Iaizzo, Dr. Jake Hutch, Tinen Iles, the data will be stored securely in Mayo B172 or with the anesthesiologist. The data will be stored from the automated TOF and the manual TOF performed in Mayo B172 or with the anesthesiologist.

References:

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy subjects (adults) admitted for surgical procedures.

Exclusion Criteria:

* Under 18 years of age or over 80 years of age, anesthetic paradigm does not include NMBAs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Quantitative Amplitude of Force in the Neuromuscular Block Aid compared to the Qualitative Standard of Care Observations | 2 years
  FDA clinical trials have utilized ~100-400 patients to determine the relative safety and efficacy of a medical device. Direct comparison of the devices qualitative evaluation of scoring from the administering anesthesiologist will be used for the final analysis.
  A peripheral nerve stimulator, used to elicit a train-of-four (TOF) response, allows the assessment of neuromuscular blockade. Subjectively they determine the relative depth by visualizing TOF responses.If the first and last stimulus in a TOF elicit no force, this indicates blockade, or if the TOF has equal amplitudes, this indicates no blockade or reversal. Return of muscle force is required before the patient can be extubated.
  Current peripheral nerve stimulators rely on visual subjective analysis of relative contractions, whereas our investigational device will provide a quantitative assessment of the amplitude of the muscle contraction in grams and percent amplitudes of measured forces relative to the first stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Iaizzo, PhD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hong JB, Iaizzo PA. Force assessment of the stimulated arm flexors: quantification of contractile properties. J Med Eng Technol. 2002 Jan-Feb;26(1):28-35. doi: 10.1080/03091900110099558. PMID 11924844
- [Result] Hong J, Falkenberg JH, Iaizzo PA. Stimulated muscle force assessment of the sternocleidomastoid muscle in humans. J Med Eng Technol. 2005 Mar-Apr;29(2):82-9. doi: 10.1080/03091900412331271158. PMID 15804857